CLINICAL TRIAL: NCT04793503
Title: Biting Force and Chewing Efficiency of Conventional and CAD/CAM Complete Dentures: A Cross-over Study
Brief Title: Biting Force and Chewing Efficiency of Complete Dentures.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Nourhan Ahmed Ragheb, lecturer of prosthodontics, Kafrelsheikh University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: KD/07/21
Record Dates: First submitted 2021-01-24; First posted 2021-03-11 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Biting; Chewing Problem
Keywords: complete denture; Biting force; chewing efficiency; CAD/CAM
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Intervention Model Description: To reduce the effect of order of treatment on MBF, were successively given the following prosthesis i) complete dentures fabricated by the conventional technique ii) 3D printed complete dentures iii) milled complete dentures in a random order.
Who Masked: Participant
Masking Description: the patient doesn't recognise the type of complete denture that he use
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- conventional complete denture (Active Comparator): the patients receive conventional complete denture constructed from heat cure acrylic resin
  Interventions: Other: conventional complete denture
- CADCAM 3D printed denture (Active Comparator): the patients receiveCADCAM 3D printed denture constructed by using printing machine
  Interventions: Other: CADCAM 3D printed denture
- CAD/CAM milled denture (Active Comparator): the patients receiveCADCAM 3D printed denture constructed by using milling machine
  Interventions: Other: CAD/CAM milled denture

INTERVENTIONS:
Other: conventional complete denture — the complete denture constructed by packing technique
  Arms: conventional complete denture
Other: CADCAM 3D printed denture — The files from the laser-scan will be translated into stereolithography (STL) files and the CDs are virtually designed in ExoCad software
  Arms: CADCAM 3D printed denture
Other: CAD/CAM milled denture — Once the complete denture has been virtually designed in CAD software (ExoCad software) a preview will be sent for evaluation using 3D viewing software
  Arms: CAD/CAM milled denture

SUMMARY:
The aim of this study was to compare the MBF and chewing efficiency of complete denture bases fabricated by conventional, 3D printing and milling techniques. The research hypothesis was that, there are no signiﬁcant differences in MBF and chewing efﬁciency in complete dentures fabricated by the three methods.

DETAILED DESCRIPTION:
Participant selection and treatment This study will include a clinical experiment with a cross-over clinical trial design. For this study, 27completely edentulous participants with age range of 50-65 were selected from the outpatient clinic of the Removable Prosthodontic Department, Faculty of dentistry, Kafr Elsheikh University, Egypt. All participants had Angle class I jaw relation maxillomandibular relationship, normal alveolar ridge volume, no temporomandibular joint disorders, no heart disease, and no systemic diseases that affect the complete denture treatment procedures.

To reduce the effect of order of treatment on MBF, were successively given the following prosthesis i) complete dentures fabricated by the conventional technique ii) 3D printed complete dentures iii) milled complete dentures in a random order.

Construction of the CADCAM 3D printed denture The same steps of the conventional technique will be performed till the adjustment of occlusion rims then in the dental laboratory, the maxillary and mandibular definitive casts and the occlusal rims will be prepared for scanning with scan spray. Scanning will be performed with an optical 3D scanner . The files from the laser-scan will be translated into stereolithography (STL) files and the CDs are virtually designed in ExoCad software. After minor modifications in the positions of teeth were made, fabrication of the dentures will be approved and the digital denture base will be fabricated using 3D printing technique from Dental Pink resin

Construction of the CAD/CAM milled denture Once the complete denture has been virtually designed in CAD software (ExoCad software) a preview will be sent for evaluation using 3D viewing software. After minor modifications in the positions of teeth were made, fabrication of the dentures will be approved. The digital denture will be fabricated by the command software of the milling machine (ExoCad 5x milling machine) from prepolymerized resin acrylic pucks and the teeth (TSM Acetal Dental) were milled into template .After that the denture will be finished and polished according to the traditional procedures For all groups, after placement, clinical evaluations of the fit, retention, stability, occlusal relationship, esthetics, and phonetics were performed. Assessment of the occlusion was made with articulating paper, chairside adjustments were made and premature contacts were corrected. The patient was given a proper program for denture insertion and oral hygiene measures.

Assessment of biting force

* This will be made by using a custom-made device composed of Flexiforce A 301® force sensor and Arduino microcontroller with a crystal display. The sensor is calibrated by known weight object for several times, and the sensor is covered by 3 mm layer of putty rubber base material.
* Readings will be performed at 1 week, 1 month and 3 months follow-up periods. Assessment of chewing efficiency The chewing efﬁciency will be evaluated according to the procedure described by Schimmel et al. (2007) using a chewing gum. Specimens will be prepared from two colored gums one with the ﬂavor "Sour Berry" (white color) and the other with the ﬂavor "Fancy Fruit" (orange color). Two strips of a standard size (30 9 18 9 3 mm) will be cut from each gum and manually stuck together. Patients will be instructed to chew ﬁve samples of gum on their preferred chewing side for 5, 10, 20, 30 and 50 cycles, respectively. Between the different tests, an interval of at least 1 min will be imposed to reduce the effect of fatigue. The total duration of the experiments was approximately 8 min.

After chewing, the samples will be then spat into transparent plastic bags, which The samples will be then scanned from both sides with a of resolution 500 dots per inch. The numbers of selected pixels will be recorded from the histogram for each side, and mean of those ﬁgures will be calculated. To assess the reproducibility of chewing, the subjects will be available to repeat the experiments on a different day.

ELIGIBILITY:
Inclusion Criteria:

* Angle class I jaw relation maxillomandibular relationship
* Normal alveolar ridge volume
* No temporomandibular joint disorders
* No heart disease
* No systemic diseases that affect the complete denture treatment procedures

Exclusion Criteria:

* Abnormal jaw relation
* TMJ disorders
* Any systemic disease interfering with complete denture treatment

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-12-02 (Actual)

PRIMARY OUTCOMES:
biting force | Readings will be performed baseline 1 week after denture insertion then 1 month after denture insertion then 3 months after denture insertion.
  - This is done custom-made device composed of Flexiforce A 301® force sensor and Arduino microcontroller with a crystal display. The sensor is calibrated by known weight object for several times, and the sensor is covered by 3 mm layer of putty rubber base material.
  • The device was placed between the upper and lower first molar. The patient then was instructed to bite as hard as possible for a period of 3 s three times in succession, with at least 20 s of resting between each bite. The readings were recorded, and the average bite force was calculated

SECONDARY OUTCOMES:
chewing efficiency | 3 months after denture insertion
  Specimens will be prepared from two colored gums one with the ﬂavor "Sour Berry" (white color) and the other with the ﬂavor "Fancy Fruit" (orange color). Two strips of a standard size (30 9 18 9 3 mm) will be cut from each gum and manually stuck together.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry , Kafr El Shiekh University, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
mean and standard deviation for each outcome in each group
Supporting Information: Study Protocol